CLINICAL TRIAL: NCT00251108
Title: The Efficacy of a Supervised Fitness Centre-Based Exercise Programme Compared to an Unsupervised Home-Based Exercise Programme on Improving Fitness and Psychosocial Outcomes in a Traumatic Brain Injured Population
Brief Title: Fitness Training After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sydney South West Area Health Service (Other Government)
Collaborators: Motor Accidents Authority of NSW (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/052; 02/040
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Craniocerebral Trauma
Keywords: 'traumatic brain injury'; 'head injury'; 'brain injuries'; 'exercise therapy'; 'physical fitness'
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Brain Injuries

INTERVENTIONS:
Procedure: Cardiorespiratory fitness training

SUMMARY:
The aim of this project is to compare the efficacy of two different fitness exercise programmes on improving fitness and psychosocial functioning in a traumatic brain injured population. We hypothesize that a supervised fitness-centre based exercise programme, compared to an unsupervised home-based exercise programme will show significant improvements in cardiorespiratory fitness, depression and community integration.

DETAILED DESCRIPTION:
The objective of this project is to compare a three-month supervised fitness centre-based exercise programme to a 3-month unsupervised home-based exercise programme on discharge from inpatient rehabilitation on improving cardiorespiratory fitness and psychosocial functioning in a traumatic brain injured population. We plan to carry out a multi-centre, assessor blinded, randomised controlled trial with a parallel group design to compare the two interventions. We hypothesise that the supervised fitness-centre based programme will provide significantly better outcomes, and that these gains will not only be evident on completion of the programme, but will be maintained on follow-up, thereby demonstrating that investment in a supervised exercise programme can provide beneficial long-term effects.

ELIGIBILITY:
Inclusion Criteria:Patients who have sustained a traumatic brain injury who have completed their inpatient rehabilitation at either of the three Sydney Metropolitan Brain Injury Units (Liverpool, Ryde or Westmead) will be included in this study if they:

* have sustained a very severe or extremely severe traumatic brain injury
* have had a hospital admission of > 1 month
* are able to walk independently at > 1 m/s on discharge
* are able to commit 3 hours per week to a fitness programme
* live within the area serviced by the 3 units

Exclusion Criteria:

* have a concurrent medical condition for which moderate to high intensity exercise is contraindicated
* are still in Posttraumatic Amnesia (PTA)
* have cognitive or language problems that affect their ability to understand verbal instructions
* have behaviour problems not suitable for a fitness centre environment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-10; Study Completion 2007-03

PRIMARY OUTCOMES:
Measure of Cardiorespiratory fitness:Modified 20 metre Walk/Run Shuttle Test:

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales (DASS)
Profile of Moods Scale (POMS)
BICRO-39
Sydney Psychosocial Reintegration Scale (SPRS)
Body Mass Index (BMI)
Rate of Perceived Exertion (RPE)
Hip to Waist ratio

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Hassett, MHSc, Principal Investigator — Brain Injury Rehabilitation Unit, Liverpool Health Service, SSWAHS; Robyn Tate, PhD, Principal Investigator — Rehabilitation Studies Unit, Royal Rehabilitation Centre Sydney; Anne M Moseley, PhD, Principal Investigator — University of Sydney; Alison R Harmer, PhD, Principal Investigator — University of Sydney
Locations (3):
- Australia (3):
  - Brain Injury Rehabilitation Unit, Royal Rehabilitation Centre Sydney, Sydney, New South Wales
  - Brain Injury Rehabilitation Unit, Liverpool Health Service, Sydney, New South Wales
  - Brain Injury Rehabilitation Unit, Westmead Hospital, Sydney, New South Wales